CLINICAL TRIAL: NCT03574220
Title: A Pilot Study of Adjuvant Pembrolizumab After Lung Stereotactic Body Radiotherapy (SBRT) for Medically Inoperable Early Stage Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Pembrolizumab After Lung SBRT for Medically Inoperable Early Stage Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No accrual - closed by PRMC
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7516
Record Dates: First submitted 2018-06-20; First posted 2018-06-29 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Non Small Cell Lung Cancer
Keywords: pembrolizumab; radiotherapy; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Stereotactic Body Radiotherapy (Experimental): Lung SBRT 50 Grays (Gy) in 5 fractions over 5-14 days, or 60 Gy in 3 fractions over 8-15 days.
  Adjuvant Therapy:
  Pembrolizumab 200mg IV every 21 days for 6 months
  Interventions: Drug: Pembrolizumab; Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — 200mg IV every 21 days over 6 months
  Other Names: Keytruda
Radiation: Stereotactic body radiotherapy — 50 Grays (Gy) in 5 fractions over 5-14 days, or 60 Gy in 3 fractions over 8-14 days

SUMMARY:
The purpose of this study is to see whether patients who have early stage NSCLC bigger than a certain size might benefit from receiving additional medicinal drug to treat their cancer after the SBRT Surgeons and radiation doctors have understood for some time that the chances of cancer showing up in areas outside the chest are higher for patients with tumors bigger than 3 cm, (about 1 ¼ inches). However, it is not routine to offer chemotherapy or drug treatments after radiation or surgery for lung cancer for patients with early stage lung cancer. This is because giving extra treatment in the form of chemotherapy has not shown to help patients live longer. There has been reluctance to offer additional treatments, especially chemotherapy, to patients with lung cancer who could not have surgery because of their medical issues. Even if these patients were felt to be at a higher risk of their cancer coming back, there is hesitation because the treatments can be difficult to tolerate in frail patients.

Recently, there have been very important advances in the kinds of drug therapy that are used for lung cancer patients. These kinds of drugs are called immunotherapy since they work with the body's immune system to fight the cancer. These drugs have been shown to make patients with advanced, incurable lung cancer, live longer and also to be very safe with very limited side effects. Because of these favorable characteristics, cancer specialists are interested in using these drugs for patients with curable cancer and for patients who may be too fragile for traditional chemotherapy. In this way, patients who get SBRT are already known to be fragile so cancer doctors are interested in now studying this kind of drug in SBRT patients to see if it can make patients with large tumors do better. The idea of the study then is that the patient would receive their standard SBRT and if their tumor is of a certain size that makes the risk of the cancer showing up outside the chest higher than routine, they would be considered for getting the immunotherapy drug.

Pembrolizumab is an investigational drug (also known as Keytruda), which has been approved by the FDA for use in certain types of skin cancer (melanoma), and for use in certain types of head and neck cancer. However, it has not been approved for use in other cancers such as newly diagnosed early stage NSCLC. It is FDA approved for advanced NSCLC, that is people who have already had some chemotherapy and their disease has worsened. Pembrolizumab is a monoclonal antibody that binds to the surface of some cells of the immune system and activates them against cancer cells. It is not chemotherapy.

DETAILED DESCRIPTION:
The primary objective of this pilot safety study is to determine the tolerability and feasibility of administering pembrolizumab in the adjuvant setting following completion of definitive SBRT to the lung for patients with medically inoperable early stage NSCLC with tumors greater than 3 cm in diameter

Secondary Objectives

1. Distant metastases free survival (DMFS)
2. Disease Free Survival (DFS)
3. Overall survival (OS)

Study design including dose escalation / cohorts

This is an open-label, single arm feasibility study of lung SBRT followed 2 to 4 weeks after completion by the addition of pembrolizumab.

Eligible patients will have biopsy-confirmed T1b-T3N0M0 (stage IA-IIB) non-small cell lung cancer (adenocarcinoma, squamous cell carcinoma, or large cell/NSCLC NOS), performance status 0-2, deemed medically inoperable by a thoracic surgeon or pulmonologist, and no contraindications to pembrolizumab.

The primary endpoint for this study is safety and feasibility. For the first stage of this study, 8 patients will be enrolled. If >7 of the initial 8 patients complete the therapy without experiencing a Grade >3 pulmonary toxicity or any Grade >4 toxicity, an additional 7 patients will be enrolled for a total of 15 patients. If >2 of the original 8 patients (>25%) experience a Grade >3 pulmonary toxicity or any Grade >4 toxicity the trial will be closed and the study therapy will be considered too toxic. If >4 of 15 patients (>26.7%) experience a Grade >3 pulmonary toxicity or any Grade >4 toxicity, the study drug regimen will be deemed too toxic and unsafe. If >12 out of 15 patients complete the study without experiencing a Grade >3 pulmonary toxicity or any Grade >4 toxicity, the study drug regimen will be considered safe and feasible for further study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed T1b-T3N0M0 (stage IA-IIB) NSCLC, which have been judged to be medically inoperable and will have undergone a course of lung SBRT will be enrolled in this trial. Eligible patients who will have completed lung SBRT will have had appropriate staging studies identifying them as specific subsets of American Joint Committee on Cancer (AJCC) 7th edition stage I or stage II based on only one of the following combinations of primary tumor, regional nodes, metastasis (TNM) staging using size criteria:

  * A. T2a (>3cm, < 5cm) N0 M0, Stage IB
  * B. T2b (>5 cm, < 7cm) N0 M0, Stage IIA
  * C. T3 (>7cm) N0 M0, Stage IIB

In order to be eligible for participation in this trial, the subject must:

* Be willing and able to provide written informed consent/assent for the trial.
* Have measurable or unmeasurable disease based on RECIST 1.1.
* Be willing to provide archival tissue from a tumor lesion.
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* All screening labs should be performed within 10 days of treatment initiation.

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9g/dL or ≥5.6mmol/L without transfusion or erythropoietin dependency (within 7 days of assessment
  * Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or measured or calculated creatinine clearance ≥ 60 mL/min for subjects with creatinine levels > 1.5 times ULN
  * Serum total bilirubin ≤ 1.5 times ULN or direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
  * aspartate aminotransferase (AST) (SGOT) and Alanine transaminase (ALT) (SGPT) ≤ 2.5 times ULN or ≤ 5 times ULN for subjects with liver metastases
  * Albumin ≥ 2.5mg/dL
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception - Contraception, for the course of the study through 120 days after the last dose of study medication.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

- Male subjects of childbearing potential must agree to use an adequate method of contraception - Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

* Has received lung SBRT for stage IA disease, or for any T2 primary tumors involving the main bronchus, 2 cm of more distal to the carina; or with associated with atelectasis that extends to the hilar region; or for any T3 tumors that invade the chest wall, mediastinal pleura, diaphragm, phrenic nerve, parietal pericardium, tumor or the main bronchus less than 2 cm distal to the carina; atelectasis of the entire lung; or with separate tumor nodule(s) in the same lobe.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known history of active Bacillus Tuberculosis (TB).
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has had any prior chemotherapy or targeted small molecule therapy for the currently diagnosed cancer.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has known history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (HCV).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-03-21 (Actual)

PRIMARY OUTCOMES:
Percent of patients tolerant to study drug | Up to 12 months
  <60% of patients being able to complete the scheduled doses of study drug without experiencing a Grade >3 pulmonary toxicity or any Grade >4 toxicity. Good tolerability had been defined as >90% of patients being able to complete the scheduled doses of study drug without experiencing a Grade >3 pulmonary toxicity or any Grade >4 toxicity.

SECONDARY OUTCOMES:
Duration of Distant metastases free survival (DMFS) | Up to 5 years
  DMFS is defined as the time from initiation of study drug post-SBRT, until the first documented, confirmed distant-only [non local, non-regional nodal] progression of disease. DMFS will be measured and reported from the initiation of SBRT.
Duration of Disease Free Survival | Up to 5 years
  DFS is defined as the time from initiation of study drug post-SBRT that the patient survives without any signs or symptoms of that cancer. DFS will also be measured and reported from the initiation of SBRT.
Duration of Overall Survival | Up to 5 years
  OS will be measure from the initiation of SBRT until death.
Duration of Local control | Up to 5 years
  For the purpose of the study, local control will be defined as a complete response, partial response, or stable disease within the planning target volume. The duration of local control will be measured from the time of SBRT initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Videtic, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center